CLINICAL TRIAL: NCT00162006
Title: Prospective Open-Label Study of the Efficacy and Safety of Immune Globulin Intravenous (Human), 10% TVR Solution in Adult Subjects With Chronic Idiopathic Thrombocytopenic Purpura
Brief Title: Efficacy and Safety Study of a 10% Triple Virally Reduced Intravenous Immune Globulin Solution in Adult Subjects With Chronic Idiopathic Thrombocytopenic Purpura
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160002
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Immune Thrombocytopenic Purpura (ITP)
Keywords: Chronic idiopathic thrombocytopenic purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — gamma-Globulins

INTERVENTIONS:
Drug: Immune Globulin Intravenous (Human), 10% Triple Virally Reduced Solution

SUMMARY:
The purpose of this study is to evaluate whether Immune Globulin Intravenous (Human), 10% TVR (Triple Virally Reduced) Solution is an effective and safe treatment in patients with chronic idiopathic thrombocytopenic purpura.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 and <= 65 years
* ITP diagnosed at least 6 months prior to study entry by history, physical exam, blood count and blood smear
* Baseline platelet count of <= 20 x 10 to the 9th/L determined prior to administration of the study drug on the day of the first infusion
* No IVIG treatment for ITP during the two weeks prior to the first infusion of the study drug
* For females of child bearing potential, use of adequate birth control measures during study participation
* Written informed consent

Exclusion Criteria:

* Serum values of ALT, AST, alkaline phosphatase, and total bilirubin exceeding 2.5 times the upper limit of normal at screening
* Renal dysfunction defined as serum creatinine greater than or equal to 2 mg/dL at screening
* Underlying other autoimmune or lymphoproliferative disorder
* Uncontrolled hypertension
* Cardiac insufficiency NYHA III and IV, coronary heart disease (CHD) NYHA III and IV
* Malignancy or history of malignancy
* Documented selective IgA deficiency (<= 10 mg/dL)
* Treatment with another investigational drug in the four weeks prior to study entry or current treatment with another investigational product
* History of severe adverse reactions to blood and/or blood products
* Pregnancy or lactation
* Positivity for HIV, or HCV antibodies, or HBsAg
* History of unresponsiveness to IVIG defined as a peak increment in platelet count <= 20,000/µL coincident with the last IVIG treatment course prior to study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-01-13 (Actual); Primary Completion 2003-12-03 (Actual); Study Completion 2003-12-03 (Actual)

PRIMARY OUTCOMES:
Subjects Who Qualify As Treatment Responders | Baseline thru Day 15 post treatment
  Subjects who i) had at least one platelet count of ≥50 x 109/L prior to Day 15 and ii) did not require a booster dose prior to Day 15, where Day 15 refers to the fifteenth day after initiation of treatment (Day 1). Otherwise, the subject is a non-responder.

SECONDARY OUTCOMES:
Time to achieve a platelet count > 50 x 109/L | Screening visit
Time to achieve a platelet count > 50 x 109/L | Day 1 (initiation of treatment)
Time to achieve a platelet count > 50 x 109/L | Day 2
Time to achieve a platelet count > 50 x 109/L | Day 5
Time to achieve a platelet count > 50 x 109/L | Day 8
Time to achieve a platelet count > 50 x 109/L | Day 11
Time to achieve a platelet count > 50 x 109/L | Day 22
Time to achieve a platelet count > 50 x 109/L | Day 15
Time to achieve a platelet count > 50 x 109/L | Day 29 (study termination visit)
Duration of platelet response | Screening visit
Duration of platelet response | Day 1 (initiation visit)
Duration of platelet response | Day 2
Duration of platelet response | Day 5
Duration of platelet response | Day 8
Duration of platelet response | Day 11
Duration of platelet response | Day 15
Duration of platelet response | Day 22
Duration of platelet response | Day 29 (study termination visit)
Maximum Platelet Count | Screening visit
Maximum Platelet Count | Day 1 (initiation visit)
Maximum Platelet Count | Day 2
Maximum Platelet Count | Day 5
Maximum Platelet Count | Day 8
Maximum Platelet Count | Day 11
Maximum Platelet Count | Day 15
Maximum Platelet Count | Day 22
Maximum Platelet Count | Day 29 (study termination visit)
Number of Adverse Experiences | Throughout the study period of approximately 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- Czechia (4):
  - Brno
  - Hradec Králové
  - Olomouc
  - Prague
- Germany (2):
  - Giessen
  - Halle
- Hungary (4):
  - Debrecen
  - Győr
  - Szeged
  - Szombathely
- Lodz, Poland